CLINICAL TRIAL: NCT01938508
Title: Bioequivalence Study Between Two Medications for the Oral Administration of 100 mg of Minocycline in Oral Solids in Healthy Volunteers.
Brief Title: Minocycline Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CECYC (Center of Scientific and Clinical Studies, CRO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200611
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Skin Diseases
Keywords: dermatitis; Minocycline; bioavailability
MeSH Terms: conditions — Skin Diseases; Dermatitis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Minocycline 100 mg capsules Darier SA Dermatological Laboratories de CV (Micromycin ®).
  Interventions: Drug: Minocycline
- Reference (Experimental): Minocycline 100 mg capsules (Micocin ®) Marketed and distributed by Triax Pharmaceuticals
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — minocycline hydrochloride capsules in microgranules equivalent to 100 mg of minocycline

SUMMARY:
This study compared the bioavailability of two formulations 100 mg (one capsule or other respectively) of each one of the products, of Minocycline, under fasting conditions, in healthy Mexican volunteers of both sexes. The single dose study under fasting (10 hours prior to study) conditions, cross, with two treatments, two periods, two sequences (2x2) randomized sequence, balanced, and with a washout period of at least 7 days between each dose, in 24 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 55 years, of both genders.
* Subjects who are in good health, based on the results of a complete medical history, valid for 6 months prior to baseline.
* Subjects with laboratory studies, liver transaminases, hepatitis B test and C, HIV and Venereal Disease Research Laboratory (VDRL). These laboratory studies have been issued within 6 months prior to the start of this study.
* Subjects who have 12-lead ECG no more than six months prior to baseline and this should be normal or normal physiologic variants.
* Subjects that have a normal chest radiograph or physiologically normal anatomic variants.
* Subjects with negative result in urine drug tests.
* Subjects with negative test alcoholometry.
* Female subjects with urine pregnancy test negative.
* Subjects with a Body Mass Index (BMI) ranging from 19 to 26.5 kg/m2.
* Subjects with laboratory results within the reference values or to +/- 10%. And if you have isolated abnormality above 10% is considered low clinical relevance criterion of Principal Investigator and indicate the relevance or otherwise of voluntary participation, as long as they ensure the safety of volunteers.
* Subjects with vital signs diastolic pressure between 50 and 89 mmHg and between 90 and 139 mmHg for systolic, pulse rate between 55 and 100 beats per minute, respiratory rate of 12-24 breaths per minute and a temperature of 35.0 to 37.5 ° C.
* Nonsmokers or smokers who have not smoked at least 10 hours before the start of the study.
* Without alcohol intake for 48 hours prior to study drug administration.
* Subjects signed informed consent, having informed the potential risks and benefits of participation, and their willingness and availability to participate in the full study, may leave the study at the time they so choose.
* Female participants must not be pregnant or breast-feeding, plus those who are sexually active should have a method of birth control to prevent pregnancy during the investigation considered the following secure methods (Male condom combined with a vaginal spermicide (Foam, gel, film, cream, or suppository, combined with a male condom female diaphragm, either with or without a vaginal spermicide, intrauterine device and also provide you with a list of other contraceptive methods in order that you do not become pregnant during the investigation).
* Prior to joining the first period sign a commitment letter no pregnancy.

Exclusion Criteria:

* Subjects with a history of hypersensitivity to the study drug or any other drugs belonging to the group of study drug.
* Subjects with a history of cardiovascular disease, renal, hepatic, metabolic, gastrointestinal, neurological, endocrine, hematopoietic, psychiatric or other organic abnormalities.
* Subjects requiring any other medications that interfere with the quantification and / or kinetic study drug.
* Subjects exposed to agents known as inducers or inhibitors of hepatic enzyme systems.
* Subjects who had taken potentially toxic drugs within 30 days before the start of the study.
* Subjects who have taken any drug within 14 days or 7 half-lives before the start of the study.
* Subjects who were hospitalized for any reason or were seriously ill within 60 days before the study.
* Subjects who have received an investigational drug within 60 days before the start of the study.
* Subjects who have donated or lost 450 mL or more of blood within 45 days prior to baseline.
* Subjects with a recent history of drug abuse, including alcohol.
* Female subjects with a positive pregnancy test in urine.
* Subjects who consumed food or beverages that interact pharmacologically with the study drug (particularly those that are known sources of xanthines: caffeine, cola drinks, theobromine, and theophylline in the 10 hours before the test.
* Subjects with grapefruit juice consumption in the 10 hours before the test.
* Subjects with inability to understand or unwilling to sign the consent form.
* Subjects who are discharged from the database by COFEPRIS are participating in another study of bioequivalence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bioavailability as assessed by composite of PK parameters. | The samples were collected for each period to 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, 36.0, 48.0 and 72.0 hours after administration
  The following pharmacokinetic (PK) parameters will assessed maximum observed concentration (Cmax), Area under the concentration time curve from time zero (pre-dose) to last common time of quantifiable concentration within a subject across all treatments (AUC0-t) and Area under the concentration time curve from time zero (pre-dose) extrapolated to infinite time (AUC0-inf).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico